CLINICAL TRIAL: NCT01713816
Title: Noninvasive Antioxidant Quantification in the Human Brain Under Oxidative Stress
Brief Title: Human Brain Antioxidants During Oxidative Stress
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1208M18321; R01AG039396 (NIH)
Record Dates: First submitted 2012-10-22; First posted 2012-10-25 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Oxidative Stress; Alzheimer's Disease; Aging
Keywords: Glutathione; Ascorbate; Alzheimer's disease; Aging; Magnetic Resonance Spectroscopy
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elderly control: Healthy elderly subjects age and gender matched to the AD cohort, predominantly male

SUMMARY:
Antioxidants are important for having a good memory and for smart thinking when people get old, and that is important for everyone's quality of life. This research will find out if normal aging and Alzheimer's disease use up brain antioxidants. It will develop a new imaging tool that can help doctors to stop cognitive decline.

DETAILED DESCRIPTION:
The objective of this proposal is to advance the mission of improving the health and well-being of older Americans by augmenting ongoing dementia prevention and treatment initiatives. It undertakes research on dementia associated with both normal aging and AD. A new scientist will develop a novel and powerful human brain antioxidant assay using state-of-the art instrumentation. The approach will be translated to the clinical environment so that it can be disseminated for use with new research. Specifically, the concentrations of two important antioxidants, ascorbate (Asc) and glutathione (GSH) will be measured noninvasively in the human brain. One aim is to measure whether a recent finding of lower brain GSH concentration in the occipital cortex of cognitively normal elder subjects is also found in the posterior cingulate cortex, and whether human brain Asc homeostasis persists in both brain regions. A complementary specific aim is to determine whether lower brain GSH concentration also occurs under the oxidative stress associated with Alzheimer's disease (AD). At the same time, data measured in subjects with AD have potential to advance this powerful new technology toward discovering an early stage biomarker. A sub aim is to make this technology available to a wide range of physicians and investigators. As such, data processing will be fully automated using commercially available software. This novel noninvasive technology facilitates a paradigm shift from systemic assays to quantifying antioxidants directly in the affected brain region. The approach will take advantage of state of the art 7 T instrumentation while developing analogous methods on a clinical 3 T scanner. The process of optimizing magnetic resonance spectroscopy (MRS) for quantification of brain Asc and GSH concentrations necessitated reliable quantification of an extensive neurochemical profile (i.e. 19 brain metabolites), which includes the four compounds that are typically observed. Spectra acquired in stimulated echo acquisition mode (STEAM) will be de-convolved quantitatively into contributions from the metabolites that contribute discernable resonances using a linear combination model approach (LCModel). Reliable quantification of brain GSH and Asc concentrations will first be achieved using ultra high field MRS with multiple transmit coil technology and accompanying radiofrequency (B1) shimming, then translated to a lower field clinical platform. Successful completion will determine whether low brain glutathione concentration is widespread in the elder human brain and whether this difference is exacerbated by AD.

ELIGIBILITY:
Inclusion Criteria:

Age and gender match to AD patients: age range 65-89:

note that we anticipate that our patients will be predominantly male, so we are NOT likely to enroll females for this portion of the study

Exclusion Criteria::

Claustrophobia Implanted metal devices Pregnancy > RDA dietary supplements

≥ 5 F+V per day Smoking Depression Poor health or systemic illness Medial history of or evidence for cognitive problems Unstable medication usage Neurological problems Psychiatric disorder Substance abuse Usage of investigational drugs Inability to complete cognitive tests written in and calibrated for English speakers Inadequate vision or hearing to accommodate participation MMSE (dementia) score ≤ 26

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: All data have been accrued for the healthy aging aim, which included healthy people age 18-22 and age 70-89. To study the second aim, 23 patients with AD will be recruited from the Minneapolis, MN VA medical center. 23 age - and gender- matched controls will be recruited to study neurodegenerative disease associated demand on the antioxidant system. We do NOT currently have the resources to screen candidates with AD who are not current patients at the VA medical center in Minneapolis.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2013-06; Primary Completion 2017-06-01 (Actual); Study Completion 2018-07-24 (Actual)

PRIMARY OUTCOMES:
Antioxidant in Alzheimers | 1 year
  Occipital cortex and posterior cingulate ascorbate and glutathione concentration in young and elder patients as well as in patients with AD

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Terpstra, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States